CLINICAL TRIAL: NCT02259244
Title: Effect of the Mediterranean Diet and Hypolipemic Reduction Diet in Combination With Exercise in Obese Croatian Population- 1-year Randomized Controlled Trial
Brief Title: Effect of Mediterranean and Hypolipemic Reduction Diet in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Collaborators: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Prof. dr. sc. Velimir Božikov, Head of the Department of Endocrinology, Diabetes and Metabolism Disorders, Dubrava University Hospital, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 006-0000000-3521
Record Dates: First submitted 2014-09-23; First posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Weight Reduction Programs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mediterranean diet+physical activity (Experimental): Mediterranean diet based on 1573 kcal/day with the goal of consumption of 30 ml/day of olive oil, 56g/week of nuts, 3-4 servings/week of fish, 3 servings/day of fruits, 2-3 servings/day of vegetables, 3 servings/week legumes and white meat instead of red meat
  Interventions: Behavioral: Weight reduction program
- Hypolipemic reduction diet+physical activity (Active Comparator): Hypolipemic reduction diet based on 1287 kcal/day with the goal of consumption of 3 servings/day of fruits, 2-3 servings/day of vegetables, 3 servings/week legumes and white meat instead of red meat, non-fat or low-fat dairy products
  Interventions: Behavioral: Weight reduction program

INTERVENTIONS:
Behavioral: Weight reduction program

SUMMARY:
The purpose of this study is to evaluate the combined effect of physical activity and adherence to Mediterranean diet or Hypolipemic Reduction diet on parameters of oxidative stress in obese patients enrolled in the weight management reduction program.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m2

Exclusion Criteria:

* newly diagnosed diabetes, hypertension or cardiovascular disease
* change in antihypertensive therapy and antidiabetic therapy in the period of 3 months prior to the commencement of the study
* insulin therapy
* alcohol consumption >500 g of alcohol/week in the last year
* pregnancy or breast feeding
* use of drugs affecting weight control (eg. weight loss medication or systemic glucocorticoids)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-10; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Oxidative stress | The outcome measure is studied at baseline, 1 and 12 months

SECONDARY OUTCOMES:
Body weight (kg) | The outcome measure is studied at baseline, 1 week, 1 month, 3, 6 and 12 months
Waist circumference (cm) | The outcome measure is studied at baseline, 1 week, 1 month, 3, 6 and 12 months
Fasting glycemia | The outcome measure is studied at baseline, 1 week, 1 month, 3, 6 and 12 months
Lipid profile (HLD, LDL, TC,) | The outcome measure is studied at baseline, 1 week, 1 month, 3, 6 and 12 months
Urate | The outcome measure is studied at baseline, at 1 week, 1 month, 3, 6 and 12 months
Blood pressure (mmHg) | The outcome measure is studied at baseline, at 1 week, 1 month, 3, 6 and 12 months
Physical activity level | The outcome measure is studied at baseline, at 1 month, 3, 6 and 12 months
  IPAQ-SF for record on physical activity during 7 last 7 days.
Quality of life | The outcome measure is studied at baseline, at 1 month, 3, 6 and 12 months
  SF-36 questionnaire
Dietary intakes | The outcome measure is studied at baseline, at 1 month, 3, 6 and 12 months
  Food Frequency Questionnaire 7-day food diary